CLINICAL TRIAL: NCT00212654
Title: Controlled Study of ONO-1101 in Patients With Postoperative Tachyarrhythmias in Japan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-1101-21
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Postoperative Supraventricular Tachyarrythmia
Keywords: ONO-1101; Landiolol Hydrochloride; Postoperative; supraventricular tachyarrhythmia
MeSH Terms: interventions — landiolol

INTERVENTIONS:
Drug: ONO-1101

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ONO-1101 in postoperative supraventricular tachyarrhythmias.

ELIGIBILITY:
Inclusion Criteria:

1. 20 years or older
2. Postoperative supraventricular tachyarrhythmias
3. Within 7 days postoperatively
4. Other inclusion criteria as specified in the protocol

Exclusion Criteria:

1. Acute myocardial infarction (within 1 month after onset)
2. Severe heart failure [New York Heart Association (NYHA) functional class III or higher]
3. Atrioventricular block (grade II or higher), or sick sinus syndrome
4. Other exclusion criteria as specified in the protocol

Ages: 21 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165
Dates: Start 2001-06; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who met the heart rate reduction criteria (20% reduction from the baseline heart rate and a heart rate of <100 beats/min)

SECONDARY OUTCOMES:
Heart rate, blood pressure, rate-pressure-product and ECG

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Development Planning, Study Director — Ono Pharmaceutical Co. Ltd